CLINICAL TRIAL: NCT02930629
Title: Assessment of Residual Paralysis in Patients in the Postoperative Anaesthetic Care Unit (PACU)
Brief Title: Residual Block in Postoperative Anaesthetic Care Unit
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1607 PACU residual block; 2016/2478 (Registry Identifier: SingHealth Centralised Institutional Review Board)
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Neuromuscular Blockade
Keywords: Recovery Period, Anesthesia; Neuromuscular Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Train-of-Four (TOF) Watch — For patients, on arriving in PACU after having had muscle relaxants during general anaesthesia
  * Two ECG electrodes will be placed 4 cm apart over the path of the ulnar nerve of the wrist after cleaning the skin with alcohol swabs.
  * The TOF force transducer will be placed on the volar aspect of the thumb.
  * The TOF Watch leads will be attached to the ECG electrodes.
  * A TOF stimulus will be applied: four twitches at 2Hz (every 0.5 seconds), each twitch lasting 0.2ms, and at a current of 50 mA. As far as possible, this will be done when patients are still slightly drowsy from the effects of anaesthesia.
  * Two TOF ratio will be elicited (two sets of four twitches 15 seconds apart), and an average of the two taken

SUMMARY:
The purpose of this study is to assess the incidence of residual block in patients arriving in the Post Anaesthetic Care Unit (PACU) following surgery, and in those who have received neuromuscular blocking drugs (muscle relaxants). Residual block (decreased motor function) due to residual levels of muscle relaxants is associated with increased morbidity.

DETAILED DESCRIPTION:
This is a prospective, cross sectional study. Adult patients undergoing surgery in the main operating theatres of Singapore General Hospital and requiring general anaesthesia and muscle relaxants will be enrolled and assessed over a 4 month period.

Explanation, handing over of the Participation Information Sheet, and consent taking for the research will be taken either: In the anaesthetic Pre-operative Evaluation Clinic (PEC) which takes place on average 1-2 weeks prior to surgery itself; or On the ward, as a portion of patients are admitted as an inpatient the day before surgery. This allows patients time to consider participation into the study.

The conduct of anaesthesia before arrival in PACU is left to the discretion of the attending anaesthetist. After arrival in PACU, patients are cared for by the PACU nurse and attending anaesthetist. The PI or co-investigators of the participants will follow up patients arriving in PACU if they fit the inclusion criteria i.e. who have received muscle relaxants during their anaesthetic.

Participants will have their neuromuscular function monitored using a TOF Watch. This is a neuromuscular monitor used to assess the twitch height of muscles when stimulated by small electrical currents. Assessing neuromuscular function at all stages of anaesthesia (during anaesthesia and during recovery from anaesthesia) is the standard of care and is considered "essential" as per guidelines from the Association of Anaesthetists of Great Britain and Ireland (2015).

The following are standards of care in PACU if patients are suspected of having residual block:

1. Neuromuscular function will be assessed using clinical means (head lift and hand grip) but these are unreliable (false positives due to effects of anaesthetic agents and opioids rather than muscle relaxants)
2. Neuromuscular function assessed by either TOF count (number of twitches) or TOF ratio (any fade in height of the four twitches) as per manufacturer's guidelines. Two ECG electrodes will be placed 4 cm apart over the path of the ulnar nerve of the wrist after cleaning the skin with alcohol swabs. The TOF force transducer will be placed on the volar aspect of the thumb. The TOF Watch leads will be attached to the electrodes and a TOF stimulus will be applied: four twitches at 2Hz (every 0.5 seconds), each twitch lasting 0.2ms, and at a current of 50 milliamperes (mA).
3. Patients who have residual block will be closely monitored as per standard care in PACU, which include oxygen therapy, and monitoring (continuous ECG, respiratory rate, pulse oximetry, and 15 minutely non invasive blood pressure measurements). Those patients who have clinical signs and symptoms of residual block will be treated at the discretion of the PACU nurse and attending anaesthetic medical officer stationed in PACU

For the research study in PACU, patients will have the above (steps 1 to 3) irrespective of whether residual block is suspected.

In addition:

The TOF ratio will be measured as two sets of TOF ratio with an average of the two taken. As far as possible, the TOF will be done when patients are still slightly drowsy from the effects of anaesthesia in order to minimize any patient TOF discomfort. If there is >10% discrepancy between these two readings then two more TOF will be applied, and an average of the two closest measurement averaged. This will determine if the participant has residual block (defined at TOF<0.9).

Medical record review of data will be that from intraoperative period and PACU stay (usually one hour) and includes data already inputted into the anaesthetic charts:

1. Patient data: age, weight, BMI, American Society of Anaesthesiologists (ASA) status, list of co-morbidities
2. Surgical data: type of operation and duration
3. Anaesthetic data: type, dose and timing of muscle relaxants and reversal used; type and method of neuromuscular monitoring used
4. PACU data: time of arrival; heart rate, blood pressure, pulse oximetry and respiratory rate on admission; any adverse incidents (airway obstruction, desaturation (SpO2<95%), complaints of muscle weakness or blurred/double vision).

ELIGIBILITY:
Inclusion Criteria:

* All patients 21 years old or older, who receive neuromuscular blocking drugs (muscle relaxants) as part of their anaesthesia for surgery.

Exclusion Criteria:

* Patients who have neuromuscular disease
* Patients for whom applying train-of-four (to detect residual block) monitoring on their ulnar nerves is not possible

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients 21 years old or older, who receive neuromuscular blocking drugs (muscle relaxants) as part of their anaesthesia for surgery, and who arrive in the postoperative anaesthesia care unit.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-08-18 (Estimated); Study Completion 2017-08-18 (Estimated)

PRIMARY OUTCOMES:
Evidence of residual block (train of four <0.9) after receiving neuromuscular block for anaesthesia for surgery | Within one hour of surgery
  Train of four is measured at the adductor pollicis using TOF Watch acceleromyography

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Wong, MBBS FRCA, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Plaud B, Debaene B, Donati F, Marty J. Residual paralysis after emergence from anesthesia. Anesthesiology. 2010 Apr;112(4):1013-22. doi: 10.1097/ALN.0b013e3181cded07. No abstract available. PMID 20234315
- [Result] Brull SJ, Prielipp RC. Reversal of neuromuscular blockade: "identification friend or foe". Anesthesiology. 2015 Jun;122(6):1183-5. doi: 10.1097/ALN.0000000000000675. No abstract available. PMID 25856292